CLINICAL TRIAL: NCT04212325
Title: Evaluation of the Effectiveness of Continuous Sciatic Nerve Block in Diabetic Foot Patients
Brief Title: Efficacy of Continuous Sciatic Nerve Block in Diabetic Foot Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/401
Record Dates: First submitted 2019-12-20; First posted 2019-12-27 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Foot; Regional Anesthesia; Catheter Blockage; Wound Heal
Keywords: Diabetic foot; Sciatic nerve catheter; wound heal
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Patients who will be operated due to diabetic foot will be randomized to 3 groups with continuous sciatic nerve block (Group C), single injection sciatic nerve block (Group S)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Continuous sciatic nerve block) (Active Comparator): Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the popliteal location 1-3 cm cephalad to the sciatic bifurcation.
  Interventions: Procedure: Group C (Continuous sciatic nerve block)
- Group S (sciatic nerve block) (Active Comparator): Patients randomized to this group will receive a sciatic nerve block with the single injection at the popliteal location 1-3 cm cephalad to the sciatic bifurcation.
  Interventions: Procedure: Group S (sciatic nerve block)

INTERVENTIONS:
Procedure: Group C (Continuous sciatic nerve block) — Patients randomized to this group will receive a sciatic nerve block with the catheter tip insertion at the popliteal location 1-3 cm cephalad to the sciatic bifurcation. After Catheter placement outcome measures will be assessed.
  Arms: Group C (Continuous sciatic nerve block)
Procedure: Group S (sciatic nerve block) — Patients randomized to this group will receive a sciatic nerve block at the popliteal location 1-3 cm cephalad to the sciatic bifurcation. After single injection sciatic nerve block, outcome measures will be assessed.
  Arms: Group S (sciatic nerve block)

SUMMARY:
Patients who underwent surgery for diabetic foot were divided into three groups: sciatic nerve block (Group B), continuous nerve catheter (Group C) . Group B patients underwent preoperative popliteal ultrasound guided peripheral nerve blockage. 20 ml of 0.25% bupivacaine was administered. In Group C patients, 20% bupivacaine 20 ml was applied to the sciatic nerve with a peripheral nerve catheter and continuous infusion was started with patient controlled analgesia device.

DETAILED DESCRIPTION:
Ethics committee approval was received on 12 December 2019, numbered 19/344. The study was planned to include 90 adult patients undergoing diabetic foot surgery at Gülhane Training and Research Hospital between 12 December 2019 and February 2020. These patients were divided into three groups: sciatic nerve block (Group B), continuous nerve catheter (Group C). Group B patients underwent preoperative popliteal ultrasound guided peripheral nerve blockage. 20 ml of 0.25% bupivacaine was administered. In Group C patients, 20% bupivacaine 20 ml was applied to the sciatic nerve with a peripheral nerve catheter and continuous infusion was started with patient controlled analgesia device. Preoperative and postoperative blood flow of the popliteal and tibialis posterior arteries, pain scores of patients were evaluated with numeric rating scale and wound healing was monitored and recorded. The differences between the groups were compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* undergoing diabetic foot surgery
* spending the first postoperative night hospitalized
* age 40 years or older

Exclusion Criteria:

* inability to communicate with the investigators and hospital staff
* incarceration
* clinical neuropathy in the surgical extremity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | three days postoperatively
  Pain 0 (no pain) to 10 (worst pain imaginable), ranging from a numeric rating scale (NRS)
Arterial blood flow | Change from Baseline arterial blood flow at postoperative 15th day
  arterial tibialis posterior and arterial dorsalis pedis blood flows in the leg to be operated will be measured by doppler ultrasound
The Wagner Diabetic Foot Ulcer Grade Classification System | preoperative and postoperative 15th day
  Grade 0 - intact Skin Grade 1 - superficial ulcer of skin or subcutaneous tissue Grade 2 - ulcers extend into tendon, bone, or capsule Grade 3 - deep ulcer with osteomyelitis, or abscess Grade 4 - partial foot gangrene Grade 5 - whole foot gangrene
Analgesic consumption | during the postoperative 5th day
  total analgesic consumption during the postoperative 5th day
patient satisfaction: survey | postoperative 15th day
  This survey was scored on a scale from 0 to 6 (the number 0 is 'not satisfied' and the number 6 is 'extremely satisfied')

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B EŞKİN, M.D., Study Director — Gulhane Training and Research Hospital; Kerim B. Yılmaz, M.D., Principal Investigator — Gulhane Training and Research Hospital; Gökhan Özkan, M.D., Principal Investigator — Gulhane Training and Research Hospital; Erhan Güven, M.D., Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)